CLINICAL TRIAL: NCT07250984
Title: The Impact of Intravenous Administration of ACMP (Eptinezumab) on the Treatment of Atypical Resistant Facial Pain
Brief Title: Treatment of Atypical Resistant Facial Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Alenka Spindler-Vesel (Other)
Responsible Party: Sponsor-Investigator, Alenka Spindler-Vesel, Assoc. Prof., MD, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Other Study IDs: 0120-331/2024-2711-8
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Facial Pain
Keywords: facial pain; CGRP; intravenous ACMP
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: intravenous administration of ACMP — 30-minute infusion of 100 mg of eptinezumab, repeated after three months

SUMMARY:
Facial pain in the trigeminal nerve region, which is not a migraine headache is often very persistent and difficult to treat. Research findings suggest that, similar to the mechanisms of migraine headache, the increased concentration of calcitonin gene-related peptide (CGRP) plays an important role in the mechanisms of facial pain.

Therefore, the hypothesis is that intravenous administration of ACMP will similarly disrupt central sensitization in facial pain as it does in migraine headaches.

DETAILED DESCRIPTION:
Facial pain in the trigeminal nerve region, which is not a migraine headache (e.g., cluster headaches, trigeminal neuralgia, burning mouth syndrome), is often very persistent and difficult to treat. Despite the use of all available treatment methods is often unsuccessful. Research findings suggest that, similar to the mechanisms of migraine headache, the increased concentration of calcitonin gene-related peptide (CGRP) plays an important role in the mechanisms of facial pain. Trigeminal neuralgia has already been treated with intravenous administration of anti-CGRP monoclonal antibodies (ACMP), such as eptinezumab.

In facial pain, as in chronic migraine, both peripheral and central nervous system sensitization can occur. Central sensitization is a poorly understood biological phenomenon, although some mechanisms are known. According to current knowledge and clinical experience, CGRP likely plays a central role in central sensitization that occurs in facial pain. It is known that in chronic migraine, the concentration of CGRP in the blood is elevated.

The peripheral mechanism of sensitization is not entirely clear, but it is likely that the peripheral part of the autonomic nervous system, specifically the parasympathetic system, plays an important role. The trigeminovascular reflex, a consequence of the autonomic segmental reflex, causes peripheral sensitization. Neurogenic inflammation also occurs. Neurogenic inflammation in the meninges further sensitizes the trigeminal nerve fibers.

CGRP is important for regulating physiological processes in the human body. It is also important for the sensitization of the peripheral nervous system, which can lead to central sensitization and create a vicious cycle. Central sensitization is a source of pro-inflammatory factors that promote neurogenic inflammation.

The level of CGRP in the body depends on its production and removal from the blood. ACMP effectively inactivate CGRP, thus reducing the number of migraine episodes and their intensity. Therefore, we hypothesize that intravenous administration of ACMP will similarly disrupt central sensitization in facial pain as it does in migraine headaches. Pharmacokinetic studies with eptinezumab have shown that intravenous administration of eptinezumab leads to an immediate peak concentration of ACMP, while subcutaneous administration reaches this effect only after several days. Since the biological availability of ACMP is significantly higher in the first few days, this may lead to the most effective reduction in CGRP influx and a probable clinical reduction in facial pain.

There are some attempts in the literature to treat cluster headaches with ACMP, but there is no data available for other syndromes.

The study will take place at the Chronic Pain Treatment Department of the Clinical Department of Anesthesiology and Intensive Care at the University Medical Centre (UKC) Ljubljana and will be designed as a multidisciplinary study (neurology and anesthesiology). 10 patients with facial pain in the trigeminal nerve region who do not have a migraine headache (e.g., cluster headaches, trigeminal neuralgia, burning mouth syndrome) and who have not responded to conventional treatment approaches will be included. Each participant will be individually assessed and invited to participate in the study, followed by an explanatory conversation. After obtaining written consent, an intravenous line will be established, and standard monitoring (non-invasive blood pressure, pulse oximeter, oximetry) will be applied. A venous blood sample will be taken, followed by a 30-minute infusion of eptinezumab. A venous blood sample and the eptinezumab dose will be repeated after three months. CGRP levels, pro-inflammatory cytokines, and specific biomarkers will be monitored, before the and after three months of drug administration .

ELIGIBILITY:
Inclusion Criteria:

* facial pain

Exclusion Criteria:

* psychiatric disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pain Therapy Clinic of University Medical Centre Ljubljana
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-11-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
MIDAS score | Change of baseline levels of MIDAS at 3 and 6 months after intervention.
  The MIDAS (Migraine Disability Assessment) questionnaire measures how much migraines affect your everyday life and activities: work, household activities, school responsibilities, and leisure activities over the past 3 months.
  The total score is obtained by summing the answers to the key questions (1-5).
  1. Low scores (0-10):
     Grade I and II- mild, ittle or no disability. Migraines has no or slight imapct on activities, but overall functioning is mostly preserved. Basic treatment and lifestyle adjustments are usually sufficient.
  2. Moderate scores (11-20):
     Grade III - moderate disability. Migraines significantly interfere with work and daily life; treatment adjustment may be needed.Consideration of preventive migraine therapy is advised.
  3. High scores (21+):
  Grade IV - severe disability. Migraines greatly reduce the ability to perform daily activities; specialist evaluation Migraines significantly impair quality of life; evaluation and prevention are recommended.

SECONDARY OUTCOMES:
Biomarkers of brain injury and inflammatory response | Change of baseline levels of proinflamatory cytokines and specific biomarkers at 3 and 6 months after intervention.
  We will take blood samples for interleukin - 6, 8 and 10 (Il6, IL8, IL10), leptin, Nerve growth factor (NGF), S100 calcium-binding protein A8 (S100A8), Brain-derived neurotrophic factor (BDNF) and CGRP

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Therapy Clinic of University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided